CLINICAL TRIAL: NCT01871844
Title: A Within Group, Randomised, Phase I, Repeated Doses, Placebo and Octreotide Controlled Study in Healthy Volunteers to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Incremental Doses of ITF2984
Brief Title: ITF2984 Repeated Doses Study in Healthy Volunteers
Acronym: MAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Italfarmaco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSC/09/2984/02; 2011-003526-27 (EudraCT Number)
Record Dates: First submitted 2013-05-22; First posted 2013-06-07 (Estimated); Last update posted 2013-06-07 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Male Volunteers
MeSH Terms: interventions — BID protein, human; Octreotide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ITF2984 500 mcg/Placebo sc bid for 7 days (Experimental): TF2984 500 mcg/Placebo sc bid for 7 days
  Interventions: Drug: ITF2984 (500, 1000, 2000 mcg bid for 7 days); Drug: Placebo
- ITF2984 1000 mcg/Placebo sc bid for 7 days (Experimental): ITF2984 1000 mcg/Placebo sc bid for 7 days
  Interventions: Drug: ITF2984 (500, 1000, 2000 mcg bid for 7 days); Drug: Placebo
- ITF2984 2000 mcg/Placebo sc bid for 7 days (Experimental): ITF2984 2000 mcg/Placebo sc bid for 7 days
  Interventions: Drug: ITF2984 (500, 1000, 2000 mcg bid for 7 days); Drug: Placebo
- octreotide 50 mcg tid (Active Comparator): octreotide 50 mcg tid
  Interventions: Drug: octreotide 50 mcg tid

INTERVENTIONS:
Drug: ITF2984 (500, 1000, 2000 mcg bid for 7 days)
  Other Names: somatostatin analogue
  Arms: ITF2984 1000 mcg/Placebo sc bid for 7 days; ITF2984 2000 mcg/Placebo sc bid for 7 days; ITF2984 500 mcg/Placebo sc bid for 7 days
Drug: octreotide 50 mcg tid
  Arms: octreotide 50 mcg tid
Drug: Placebo
  Arms: ITF2984 1000 mcg/Placebo sc bid for 7 days; ITF2984 2000 mcg/Placebo sc bid for 7 days; ITF2984 500 mcg/Placebo sc bid for 7 days

SUMMARY:
This was a within group, randomised, repeated dose, placebo- and octreotide controlled study in a target population of 45 healthy male subjects. Subjects were required to attend the clinical for screening procedures between 3 and 28 days before dosing commenced. The study was conducted in 4 groups of subjects; Groups 1 to 3 were a double-blinded, randomised design, each consisting of 12 subjects. Group 4 was an open-label design and consisted of 9 subjects. There was a minimum interval of 96 h between dosing of Groups 1, 2 and 3 to allow for interim analyses of PK and safety/tolerability data for dose escalation purposes. Group 4 (the active control group) was still to proceed if the decision was taken to prematurely stop dosing with ITF2984 (somatostatin analogue) following review of the PK and safety data presented at the interim decision meeting; dosing of this group was conducted independently from Groups 1 to 3. On Days 1 to 6, subjects in Groups 1 to 3 were to receive 2 doses of investigational medicinal product (IMP) approximately 12 h apart; subjects in Group 4 were to receive 3 doses of IMP approximately 8 h apart. For all groups, subjects were scheduled to receive their final dose of IMP on the morning of Day 7.

In addition, subjects were to receive exogenous test administrations(stimulation test) on Day -1, Day 1 and Day 7 at the same time on each day (ie for Day -1, 23.5 h before the first dose of IMP, and for Days 1 and 7, 0.5 h after the first dose of IMP on the respective day). Blood samples for PD and PK analyses were taken at specified time points after each dosing.

Subjects remained on site for 10 days (ie 36 h after the final dose of IMP on Day 7) providing that discharge conditions had been met, and returned to the clinic between 5 and 10 days after the last IMP administration for a follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Caucasian male volunteers between 18 and 50 years of age, inclusive.
2. Body mass index (BMI) of 18 to 25 kg/m2 inclusive.
3. Was willing and able to communicate and participate in the entire study.
4. Had an understanding, ability and willingness to fully comply with study procedures and restrictions.
5. Was willing and able to provide written, personally signed and dated informed consent to participate in the study, in accordance with the ICH GCP Guidelines and applicable regulations, before completing any study-related procedures.
6. Agreed to comply with the applicable contraceptive requirements from admission to 90 days after the last dose.
7. Had a satisfactory medical assessment with no clinically significant or relevant abnormalities in medical history, physical examination, vital signs, ECG or laboratory evaluation (haematology, biochemistry, urinalysis) as assessed by the investigator.

Exclusion Criteria:

1. Current or recurrent disease (eg cardiovascular, respiratory, endocrine, renal, liver, GI, malignancy or other conditions) that could have affected the action, absorption or disposition of the IMP, or could have affected clinical or laboratory assessments.
2. Current or relevant previous history of physical or psychiatric illness, any medical disorder that may have required treatment or made the subject unlikely to fully complete the study, or any condition that presented undue risk from the IMP or study procedures.
3. Significant illness, as judged by the investigator, within 2 weeks of the first dose of IMP.
4. Current use (defined as use within 14 days of first IMP dose) of any medication, including prescription, over-the-counter, herbal or homeopathic preparations (other than 4 g per day of paracetamol).
5. Subjects who had received prohibited medication
6. Known or suspected intolerance or hypersensitivity to the IMP, closely related compounds or any of the stated ingredients.
7. History of alcohol or other substance abuse within the last year. A positive result for alcohol or drugs of abuse.
8. Male subjects who consumed more than 21 units of alcohol per week or 3 units per day (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine).
9. A positive human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) test.
10. Use of tobacco in any form (eg smoking or chewing) or other nicotine-containing products in any form (eg gum, patch). Ex-users had to report that they had stopped using tobacco for at least 90 days before receiving the first dose of IMP. A breath carbon monoxide (CO) reading of greater than 10 ppm at screening.
11. Donation of blood or blood products (eg plasma or platelets) of greater than 400 mL within 90 days before receiving IMP.
12. Use of another IMP within 90 days before receiving the first dose of IMP, or active enrolment in another drug or vaccine clinical study.
13. Subjects who had previously been enrolled in this study.
14. Clinically significant abnormal biochemistry, haematology or urinalysis result as judged by the investigator.
15. Presence or history of allergy requiring treatment. Hayfever was allowed as long as it was inactive.
16. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2012-01; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of ITF2984 on GH, insulin, glucagon and glucose after exogenous stimulus | 7 days
To evaluate the safety profile of repeated doses of ITF2984 | 10 days after last dose administration
  Numbers of Adverse Events
To evaluate the pharmacodynamic effects of ITF2984 on glucose, insulin, IGF-1, IGF-BP1 and IGF-BP3 | 7 days
to evaluate the effects of ITF2984 on TSH, ACTH, Cortisol, PRL, LH and FSH after exogenous stimulus | 7 days

SECONDARY OUTCOMES:
To observe the plasma concentration of ITF2984 repeated doses (500, 1000, 2000 mcg bid for 7 days) | from the first administration to 10 days after last drug administration

CONTACTS AND LOCATIONS:
Locations (2):
- Centro Ricerche Cliniche, Verona, Italy
- Quotient Clinical, Ruddington, Nottingham, United Kingdom